CLINICAL TRIAL: NCT00756002
Title: A Randomized, Double-Blind, Placebo-Controlled, Polysomnography Plus Outpatient Study to Determine the Safety and Efficacy of 4 mg Ramelteon in Adults With Chronic Insomnia
Brief Title: Safety and Efficacy Study of Ramelteon in Subjects With Chronic Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-06-TL-375-081; 2007-000403-15 (Registry Identifier: EudraCT); U1111-1115-2084 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Results first posted 2009-11-05 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Chronic Insomnia; DIMS (Disorders of Initiating and Maintaining Sleep); Disorders of Initiating and Maintaining Sleep; Insomnia Disorder Sleep Initiation Dysfunction; Transient Insomnia; Drug Therapy; Sleep Disorders, Intrinsic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Disorders, Intrinsic | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramelteon 4 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon 4 mg, tablets, orally, once daily for up to 5 weeks.
  Other Names: Rozerem™; TAK-375
  Arms: Ramelteon 4 mg QD
Drug: Placebo — Ramelteon placebo-matching tablets, orally, once daily for up to 5 weeks.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to determine the safety and efficacy of 4 mg of Ramelteon, once daily (QD), in subjects with chronic insomnia.

DETAILED DESCRIPTION:
In the western world, there are several people affected by chronic insomnia. Numerous studies estimate that 30% to 40% of the general population is affected at some time in their lives with a form of insomnia that goes on for several months, and about one third of those are described as severely affected. Daytime symptoms of insomnia include tiredness, lack of energy, difficulty concentrating and irritability. Recent epidemiologic research focusing on the quality of life has identified significant insomnia-related morbidities that relate to work productivity, health care utilization, and risk of depression. Insomnia is associated with diminished work output, absenteeism, and greater rates of accidents.

Although normal control of the sleep-wake cycle is exerted by the suprachiasmatic nucleus via melatonin receptor subtype 1 and 2 (MT1 and MT2) receptors (melatonin receptor subtype), most current pharmacologic treatments for insomnia mainly involve GABAergic (gamma-aminobutyric acid) mechanisms. Most currently prescribed sleep agents are benzodiazepine receptor agonists, which induce sleep by binding to the benzodiazepine receptor site of the gamma-aminobutyric acid-A receptor complex. Gamma-aminobutyric acid is the major inhibitory transmitter in the central nervous system, and its receptors are distributed widely throughout the brain. In addition to sleep, benzodiazepine receptor agonists can cause a wide range of ancillary effects not directly related to sleep, depending on the precise subset of gamma-aminobutyric acid-A receptors activated. These include sedative, anxiolytic, muscle-relaxant, and amnesic effects. The risk of tolerance, dependence development, and abuse potential associated with the benzodiazepine receptor agonists also may reflect effects of these drugs on the gamma-aminobutyric acid-A receptor complex.

The sleep-wake cycle results from the interaction of circadian and homeostatic mechanisms. The homeostatic mechanism refers to the accumulation of sleep load during time awake; the organism falls asleep when the sleep load is high, and the reduction of sleep load during sleep results in waking.

A circadian rhythm is superimposed on the homeostatic mechanism. Circadian rhythms are controlled by the suprachiasmatic nucleus, which emits alerting signals; this signal is believed to be attenuated by melatonin, which is produced in response to darkness. It is believed that binding of melatonin to MT1 and MT2 receptors in the suprachiasmatic nucleus inhibits firing of specific neurons, and this is thought to attenuate the alerting signal, allowing the homeostatic mechanism to express itself and promote sleep.

An agent that is selective for the MT1 and MT2 receptors would be expected to be devoid of the ancillary effects of agents that act at the gamma-aminobutyric acid-A receptor complex. It would promote sleep by specifically targeting the alerting signal in the suprachiasmatic nucleus, allowing the homeostatic mechanism to produce sleep.

Ramelteon is under global development by Takeda Pharmaceuticals as a nonscheduled sleep agent for the treatment of difficulty with sleep initiation, and is marketed under the brand name of Rozerem™ in the United States. In vitro, ramelteon demonstrates affinity and selectivity for human melatonin MT1 and MT2 receptors compared to melatonin. It also demonstrates full agonist activity in cells expressing human MT1 or MT2 receptors relative to melatonin.

In the European Union, Takeda is seeking marketing approval for the long-term treatment of transient and chronic insomnia as characterized by difficulty with sleep onset. Because most of the European clinical studies to date have used the 8 mg dose, the aim of this study is to assess the safety and efficacy of 4mg of ramelteon in a larger number of adults with chronic insomnia.

Subjects participating in this study will be required to report to a sleep laboratory and have polysomnography recordings over two consecutive nights for three sittings during a five week period. The total duration of the study is approximately 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A female subject of childbearing potential who is sexually active agrees to use adequate contraception from Screening throughout the duration of the study.
* Has a body mass index between 18 and 34, inclusive.
* Based on sleep history, the subject has had chronic insomnia for at least 3 months, as defined by the following:

  * The predominant complaint is difficulty initiating or maintaining sleep, or non-restorative sleep, for at least 3 months.
  * The sleep disturbance (or associated daytime fatigue) causes clinically significant distress or impairment in social, occupational, or other important areas of functioning.
  * The sleep disturbance does not occur exclusively during the course of narcolepsy, breathing-related sleep disorder, circadian rhythm sleep disorder, or parasomnia.
  * The disturbance does not occur exclusively during the course of another mental disorder (eg, major depressive disorder, generalized anxiety disorder, delirium).
  * The disturbance is not due to the direct physiological effects of a substance or a general medical condition.
* Based on sleep history, the subject reports a history of subjective sleep latency ≥45 minutes and a subjective total sleep time ≤6.5 hours for at least 3 months.
* Based on sleep history, the subject's habitual bedtime is between 10:00 PM and 1:00 AM.
* On at least 3 of the first 5 nights of single blind run-in placebo treatment, the subject must have an subjective sleep latency of ≥45 minutes and a subjective total sleep time of <6.5 hours.
* The difference of the average subjective sleep latency from first 3 nights of data in the first week of single-blind run-in to the average of the last 3 nights of data in the first week of single-blind run-in must be ≤30 minutes.
* The difference of the average subjective sleep latency from first 3 nights of data in the first week of single-blind run-in to the average of the last 3 nights of data in the second week of single-blind run-in must be ≤30 minutes.
* The difference of the average subjective sleep latency from first 3 nights of data in the first week of single-blind run-in to the average of the last 3 nights of data in the third week of single-blind run-in must be ≤30 minutes.
* Is willing to have a fixed bedtime and agrees to go to bed within ± 30 minutes of the habitual bedtime during the entire study, exceptions will be allowed at weekends that are not within 2 days of a polysomnography visit.
* Has consistent access to a touch-tone phone and is willing to complete all telephone questionnaires within 60 minutes of wake time each morning throughout the entire duration of the study.
* Is willing to remain in bed for at least 6.5 hours each night during the entire study.
* Based on sleep history, the subject normally uses pharmacologic assistance to sleep 0 to 4 (maximum allowable) times per week in the last 3 months. Subjects must agree to discontinue the use of all sleep aids beginning 1 week prior to the first dose of single-blind study medication and throughout the entire duration of the study.
* The subject must complete the post-sleep questionnaire morning questionnaire on at least 5 of 7 mornings for all 3 weeks of single-blind run-in.
* Has a mean latency to persistent sleep of ≥20 minutes on 2 consecutive screening nights, with neither night less than 15 minutes, via polysomnography screening assessment during the single-blind placebo run-in period.

Exclusion Criteria:

* Has a known hypersensitivity to ramelteon or related compounds, including melatonin.
* Has participated in a study involving ramelteon within 6 months of initial Screening Visit.
* Has participated in any other investigational study and/or taken any investigational drug within 30 days or 5 half-lives (whichever is longer) prior to the first night of single-blind study medication.
* Has sleep schedule changes required by employment (eg, shift worker) within 3 months prior to the first night of single-blind study medication, or has flown across greater than 3 time zones within 7 days prior to Screening.
* Has participated in a weight loss program or has substantially altered his or her exercise routine within 30 days prior to the first night of single-blind study medication.
* Has ever had a history of seizures, sleep apnea, restless leg syndrome, periodic leg movements during sleep, chronic obstructive pulmonary disease, fibromyalgia, schizophrenia, bipolar disorder, mental retardation or a cognitive disorder.
* Has a history of psychiatric disorder (including anxiety or depression) within the past 12 months.
* Has a history of drug addiction or alcohol abuse and/or regularly consumes 4 or more alcoholic drinks per day within the past 12 months, as defined in Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised.
* Has a current significant neurological (including cognitive and psychiatric disorders), hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematological, or metabolic disease, unless currently controlled and stable with protocol-allowed medication 30 days prior to the first night of single blind study medication.
* The subject uses tobacco products (including nicotine gum and patch) during nightly awakenings.
* The subject has any clinically important abnormal finding as determined by a medical history, physical examination, electrocardiogram, or clinical laboratory tests, as determined by the investigator.
* The subject is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Anxiolytics
  * Central nervous system active drugs (including herbal)
  * Hypnotics
  * Narcotic analgesics
  * Antidepressants
  * Beta-blockers
  * Anticonvulsants
  * Systemic steroids
  * Sedating H1 antihistamines
  * Respiratory stimulants
  * Muscle relaxants
  * Sedatives
  * Antipsychotics
  * Sedating decongestants
  * Kava-kava
  * St. John's wort
  * Ginkgo biloba
  * Over-the counter and prescription stimulants, diet aids and sleep aids
  * Drugs that are known or are suspected to significantly inhibit CYP450
  * Melatonin
* Has a positive urine drug screen for an illegal substance at the initial Screening Visit.
* Has a positive urine drug screen at polysomnography screening or a positive alcohol breathalyzer test at polysomnography screening or randomization.
* Exhibits a placebo response during the single-blind placebo run-in period. A placebo response is defined as having:

  * a difference in average subjective sleep latency >30 minutes from first 3 nights of data in the first week of single-blind run-in to the average of the last 3 nights of data in the first week of single-blind run-in.
  * a difference in average subjective sleep latency >30 minutes from first 3 nights of data in the first week of single-blind run-in to the average of the last 3 nights of data in the second week of single-blind run-in.
  * a difference in average subjective sleep latency >30 minutes from first 3 nights of data in the first week of single-blind run-in to the average of the last 3 nights of data in the third week of single-blind run-in.
* Has periodic leg movements during sleep with arousal index (per hour of sleep) >10 as seen on polysomnography on the first night of polysomnography screening.
* Has any additional condition(s) that in the Investigator's opinion would:

  * Affect sleep/wake function
  * Prohibit the subject from completing the study
  * Not be in the best interest of the subject to complete the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 259 (Actual)
Dates: Start 2007-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda

REFERENCES:
- See also: Rozerem Package Insert. — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 19 sites in Europe and Russia from 21 August 2007 to 28 March 2008.
Pre-assignment Details: Sleep quality was assessed by postsleep questionnaires during a 21-day placebo run-in. Subjects were enrolled in Ramelteon or Placebo once-daily (QD) treatment group.
  488 subjects entered placebo Run-in Period. 229 failed randomization criteria for entry into double-blind study medication phase of the study. 259 were randomized into the study.
Groups:
- Placebo QD: Oral Placebo was self-administered once-daily, 30 minutes prior to bedtime. The study medication consisted of identical film-coated pale orange-yellow tablets.
- Ramelteon 4 mg QD: Ramelteon 4 mg tablets, self-administered once-daily, 30 minutes prior to bedtime. Study medication consisted of identical film-coated pale orange-yellow tablets.
Period: Placebo Run-in
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Started | 488 | 0
Completed | 259 | 0
Not Completed | 229 | 0
Period: Double-Blind Treatment Period
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Started | 129 | 130
Completed | 114 | 115
Not Completed | 15 | 15
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Protocol Violation | 6 | 5
Not completed — Other | 2 | 2
Period: Placebo Run-out
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Started | 114 | 0
Completed | 114 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo QD | Ramelteon 4 mg QD | Total
Number analyzed (Participants) | 129 | 130 | 259
Age Continuous [Mean (Standard Deviation); unit: years] | 42.3 (12.28) | 41.7 (11.85) | 42.0 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 53 | 108.0
  Male | 74 | 77 | 151.0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1.0
  Black or African American | 0 | 1 | 1.0
  White | 128 | 129 | 257.0

OUTCOME MEASURES:

1. Primary Outcome: Mean Latency to Persistent Sleep Via Polysomnography (Nights 1-2).
Description: Elapsed time from the beginning of the Polysomnography recording to the onset of the first 10 minutes of continuous sleep was measured over 2 nights and the average time to sleep was calculated.
Time Frame: Nights 1-2
Population: The Full Analysis Set (FAS) population consisted of all subjects who were randomized and received at least 1 dose of double-blind study medication. Subjects were analyzed according to the treatment they were randomized to receive. The analysis was performed using the FAS and Last Observation Carried Forward (LOCF) data.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
minutes | 67.0 (2.88) | 41.7 (2.83)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; One subject did not have postsleep questionnaire data on day 2; however, had polysomnography data recorded. Analysis was based on LOCF data; Test type: Superiority or Other; p < 0.001, ANCOVA — P-values are from t-tests of the ANCOVA model for the overall treatment comparison. Statistical significance was determined at the 0.05 level; Least Squares (LS) means from ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

2. Secondary Outcome: Mean Latency to Persistent Sleep Via Polysomnography (Nights 15-16).
Description: Elapsed time from the beginning of the Polysomnography recording to the onset of the first 10 minutes of continuous sleep was measured.
Time Frame: Nights 15-16
Population: The FAS population consisted of all subjects who were randomized and received at least 1 dose of double-blind study medication. Subjects were analyzed according to the treatment they were randomized to receive. The analysis was performed using the FAS and LOCF data.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
minutes | 65.3 (3.09) | 39.2 (3.04)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS means are from ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

3. Secondary Outcome: Mean Latency to Persistent Sleep Via Polysomnography (Nights 29-30).
Description: as for outcome 2
Time Frame: Nights 29-30
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
minutes | 60.5 (2.95) | 37.2 (2.89)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS means are from ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

4. Secondary Outcome: Subjective Sleep Latency, Per Post-sleep Questionnaire (Nights 1-2).
Description: Subjective sleep latency was collected by subjects answering a post-sleep questionnaire via an interactive voice response system (IVRS) following an overnight Polysomnography in the sleep lab.
Time Frame: Nights 1-2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 129
minutes | 73.5 (2.84) | 61.5 (2.80)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS means are from ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

5. Secondary Outcome: Subjective Sleep Latency, Per Post-sleep Questionnaire (Nights 15-16).
Description: Subjective sleep latency was collected by subjects answering a post-sleep questionnaire (via IVRS) following an overnight Polysomnography in the sleep lab.
Time Frame: Nights 15-16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
minutes | 72.3 (3.29) | 55.8 (3.23)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS means are from ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

6. Secondary Outcome: Subjective Sleep Latency, Per Post-sleep Questionnaire (Nights 29-30).
Description: as for outcome 5
Time Frame: Nights 29-30
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
minutes | 72.3 (3.59) | 53.7 (3.53)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS means are from ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

7. Secondary Outcome: Subjective Sleep Latency, Per Post-sleep Questionnaire (Week 2).
Description: Subjects answered a post-sleep questionnaire via IVRS. The Subjective Sleep Latency weekly average was the mean of the daily Post-Sleep Questionnaire for the 7 nights prior to the corresponding Visit and predominantly contained data from the natural "home" setting.
Time Frame: Week 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 124 | 127
minutes | 69.9 (2.31) | 52.7 (2.27)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS means are from ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

8. Secondary Outcome: Subjective Sleep Latency, Per Post-sleep Questionnaire (Week 4).
Description: as for outcome 7
Time Frame: Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 125 | 127
minutes | 65.7 (2.22) | 51.0 (2.18)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS means are from ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

9. Secondary Outcome: Subjective Sleep Latency, Per Post-sleep Questionnaire (Week 5).
Description: as for outcome 7
Time Frame: Week 5
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 125 | 127
minutes | 67.4 (2.40) | 50.4 (2.36)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS means are from ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

10. Secondary Outcome: Total Sleep Time, Per Polysomnography (Nights 1-2).
Description: All of the minutes of Stages 1, 2, 3/4 Non Rapid Eye-Movement (NREM) and Rapid-Eye-Movement (REM) sleep, as measured by Polysomnography, are summed to determine the Total Sleep Time.
Time Frame: Nights 1-2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
minutes | 356.5 (3.76) | 381.1 (3.71)
Statistical Analysis 1: Comparison: Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS means are from ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

11. Secondary Outcome: Total Sleep Time, Per Polysomnography (Nights 15-16).
Description: All of the minutes of Stages 1, 2, 3/4 NREM and REM sleep, as measured by Polysomnography, are summed to determine the Total Sleep Time.
Time Frame: Nights 15-16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
minutes | 357.0 (4.15) | 380.3 (4.09)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS means are from ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

12. Secondary Outcome: Total Sleep Time, Per Polysomnography (Nights 29-30).
Description: as for outcome 11
Time Frame: Nights 29-30
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
minutes | 361.7 (4.19) | 386.2 (4.13)
Statistical Analysis 1: Comparison: Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS means are from ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

13. Secondary Outcome: Subjective Total Sleep Time, Per Post-sleep Questionnaire (Nights 1-2).
Description: Subjects answered a Post-Sleep Questionnaire in the sleep lab the morning following overnight Polysomnography. Subjective Total Sleep Time measured the average of the 2 mornings after each overnight Polysomnography Visit.
Time Frame: Nights 1-2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 129
minutes | 330.6 (3.45) | 347.0 (3.41)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — LS means from ANCOVA model with effects for treatment & pooled center, with Baseline as a covariate. P-values from t-tests of the ANCOVA model for the overall treatment comparison. Statistical significance was determined at the 0.05 level

14. Secondary Outcome: Subjective Total Sleep Time, Per Post-sleep Questionnaire (Nights 15-16).
Description: as for outcome 13
Time Frame: Nights 15-16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
minutes | 332.6 (4.63) | 345.9 (4.57)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.043, ANCOVA — [p-value comment as in outcome 13, analysis 1]

15. Secondary Outcome: Subjective Total Sleep Time, Per Post-sleep Questionnaire (Nights 29-30).
Description: as for outcome 13
Time Frame: Nights 29 -30
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
minutes | 335.0 (5.16) | 355.3 (5.10)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.005, ANCOVA — P-values for differences are obtained using t-tests from the ANCOVA model of the overall treatment comparison. Statistical significance was determined at the 0.05 level; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

16. Secondary Outcome: Subjective Total Sleep Time, Per Post-sleep Questionnaire (Week 2).
Description: Subjects answered a Post-Sleep Questionnaire via IVRS. The Subjective Total Sleep Time weekly average was the mean of the daily Post-Sleep Questionnaire for the 7 nights prior to the corresponding Visit and predominantly contained data from the natural "home" setting.
Time Frame: Week 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 124 | 127
minutes | 343.7 (3.65) | 357.1 (3.59)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.010, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

17. Secondary Outcome: Subjective Total Sleep Time, Per Post-sleep Questionnaire (Week 4).
Description: as for outcome 16
Time Frame: Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 125 | 127
minutes | 349.4 (3.84) | 366.7 (3.79)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

18. Secondary Outcome: Subjective Total Sleep Time, Per Post-sleep Questionnaire (Week 5).
Description: as for outcome 16
Time Frame: Week 5
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 125 | 127
minutes | 350.7 (3.90) | 366.1 (3.86)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.006, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

19. Secondary Outcome: Sleep Efficiency, Per Polysomnography (Nights 1-2).
Description: The total sleep time was divided by the total time in bed (ie, the number of minutes from the beginning of the Polysomnography recording to the end of the recording), multiplied by 100.
Time Frame: Nights 1-2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of time asleep to time in bed
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
percentage of time asleep to time in bed | 74.3 (0.78) | 79.5 (0.77)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with the Baseline value as a covariate

20. Secondary Outcome: Sleep Efficiency, Per Polysomnography (Nights 15-16).
Description: as for outcome 19
Time Frame: Nights 15-16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of time asleep to time in bed
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
percentage of time asleep to time in bed | 74.5 (0.87) | 79.4 (0.85)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with the Baseline value as a covariate

21. Secondary Outcome: Sleep Efficiency, Per Polysomnography (Nights 29-30).
Description: as for outcome 19
Time Frame: Nights 29-30
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of time asleep to time in bed
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
percentage of time asleep to time in bed | 75.6 (0.87) | 80.5 (0.86)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with the Baseline value as a covariate

22. Secondary Outcome: Subjective Sleep Quality, Per Post-sleep Questionnaire (Nights 1-2).
Description: Sleep quality obtained from the Post-Sleep Questionnaire performed in the sleep lab the morning following overnight Polysomnography. 7=Extremely Poor; 6=Very Poor; 5=Poor; 4=Fair; 3=Good; 2=Very Good; 1=Excellent.
Time Frame: Nights 1-2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
scores on a scale | 4.4 (0.06) | 4.1 (0.06)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

23. Secondary Outcome: Subjective Sleep Quality, Per Post-sleep Questionnaire (Nights 15-16).
Description: as for outcome 22
Time Frame: Nights 15-16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
scores on a scale | 4.3 (0.08) | 3.9 (0.07)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

24. Secondary Outcome: Subjective Sleep Quality, Per Post-sleep Questionnaire (Nights 29-30).
Description: Sleep quality obtained from the Post-Sleep Questionnaireperformed in the sleep lab the morning following overnight Polysomnography. 7=Extremely Poor; 6=Very Poor; 5=Poor; 4=Fair; 3=Good; 2=Very Good; 1=Excellent.
Time Frame: Nights 29-30
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
scores on a scale | 4.2 (0.08) | 3.7 (0.08)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

25. Secondary Outcome: Subjective Sleep Quality, Per Post-sleep Questionnaire (Week 2).
Description: The subjective sleep quality weekly average was the mean of the daily Post-Sleep Questionnaire for the 7 nights prior to the corresponding Visit and predominantly contained data from the natural "home" setting. 7=Extremely Poor; 6=Very Poor; 5=Poor; 4=Fair; 3=Good; 2=Very Good; 1=Excellent.
Time Frame: Week 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 124 | 127
scores on a scale | 4.2 (0.06) | 3.8 (0.06)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

26. Secondary Outcome: Subjective Sleep Quality, Per Post-sleep Questionnaire (Week 4).
Description: as for outcome 25
Time Frame: Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 125 | 127
scores on a scale | 4.1 (0.07) | 3.7 (0.07)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

27. Secondary Outcome: Subjective Sleep Quality, Per Post-sleep Questionnaire (Week 5).
Description: as for outcome 25
Time Frame: Week 5
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 125 | 127
scores on a scale | 4.1 (0.07) | 3.7 (0.07)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

28. Secondary Outcome: Wake Time After Sleep Onset, Per Polysomnography (Nights 1-2).
Description: The number of minutes in the Awake stage after the onset of persistent sleep to the end of the recording.
Time Frame: Nights 1-2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
minutes | 61.1 (2.96) | 62.2 (2.93)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.785, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

29. Secondary Outcome: Wake Time After Sleep Onset, Per Polysomnography (Nights 15-16).
Description: The number of minutes in the Awake stage after the onset of persistent sleep to the end of the recording.
Time Frame: Nights 15-16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
minutes | 62.6 (3.10) | 66.1 (3.06)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.422, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

30. Secondary Outcome: Wake Time After Sleep Onset, Per Polysomnography (Nights 29-30).
Description: The number of minutes in the Awake stage after the onset of persistent sleep to the end of the recording.
Time Frame: Nights 29-30
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
minutes | 62.4 (3.57) | 60.3 (3.52)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.665, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

31. Secondary Outcome: Subjective Wake Time After Sleep Onset, Per Post-sleep Questionnaire (Nights 1-2).
Description: Subjective Wake Time After Sleep Onset obtained from the Post-Sleep Questionnaire performed in the sleep lab the morning following overnight Polysomnography.
Time Frame: Nights 1-2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
minutes | 82.2 (3.50) | 76.3 (3.46)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.228, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

32. Secondary Outcome: Subjective Wake Time After Sleep Onset, Per Post-sleep Questionnaire (Nights 15-16).
Description: as for outcome 31
Time Frame: Nights 15-16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
minutes | 83.8 (4.01) | 74.5 (3.94)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.099, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

33. Secondary Outcome: Subjective Wake Time After Sleep Onset, Per Post-sleep Questionnaire (Nights 29-30).
Description: as for outcome 31
Time Frame: Nights 29-30
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
minutes | 81.1 (4.40) | 63.8 (4.33)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.005, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

34. Secondary Outcome: Subjective Wake Time After Sleep Onset, Per Post-sleep Questionnaire (Week 2).
Description: The Subjective Wake Time After Sleep Onset weekly average was the mean of the daily Post-Sleep Questionnaire for the 7 nights prior to the corresponding Visit and predominantly contained data from the natural "home" setting.
Time Frame: Week 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 124 | 127
minutes | 70.8 (2.68) | 59.8 (2.62)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.004, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

35. Secondary Outcome: Subjective Wake Time After Sleep Onset, Per Post-sleep Questionnaire (Week 4).
Description: as for outcome 34
Time Frame: Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 125 | 127
minutes | 65.8 (2.88) | 52.5 (2.83)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

36. Secondary Outcome: Subjective Wake Time After Sleep Onset, Per Post-sleep Questionnaire (Week 5).
Description: as for outcome 34
Time Frame: Week 5
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 125 | 127
minutes | 67.7 (2.96) | 55.7 (2.91)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.004, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

37. Secondary Outcome: Number of Awakenings After Persistent Sleep, Per Polysomnography (Nights 1-2).
Description: Number of Awakenings is defined as the number of times after the onset of persistent sleep that there is a wake entry of at least 2 epochs in duration. Each entry must be separated by Stage 2, 3/4 NREM sleep or REM sleep in order to be counted.
Time Frame: Nights 1-2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: awakenings after persistent sleep
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
awakenings after persistent sleep | 9.6 (0.30) | 10.4 (0.30)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.040, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

38. Secondary Outcome: Number of Awakenings After Persistent Sleep, Per Polysomnography (Nights 15-16).
Description: as for outcome 37
Time Frame: Nights 15-16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: awakenings after persistent sleep
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
awakenings after persistent sleep | 9.9 (0.32) | 9.7 (0.32)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.814, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

39. Secondary Outcome: Number of Awakenings After Persistent Sleep, Per Polysomnography (Nights 29-30).
Description: as for outcome 37
Time Frame: Nights 29-30
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: awakenings after persistent sleep
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
awakenings after persistent sleep | 9.8 (0.33) | 9.7 (0.33)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.929, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

40. Secondary Outcome: Subjective Number of Awakenings, Per Post-sleep Questionnaire (Nights 1-2).
Description: Subjective Number of Awakenings (the subjective measure of how many times the subject believes they awoke during the night) obtained from the Post-Sleep Questionnaire performed in the sleep lab the morning following overnight Polysomnography. The average of two nights' data is used for each subject at a visit.
Time Frame: Nights 1-2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Number of awakenings per night
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
Number of awakenings per night | 2.9 (0.12) | 2.8 (0.12)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.591, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

41. Secondary Outcome: Subjective Number of Awakenings, Per Post-sleep Questionnaire (Nights 15-16).
Description: as for outcome 40
Time Frame: Nights 15-16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Number of awakenings per night
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
Number of awakenings per night | 3.0 (0.13) | 2.6 (0.13)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.015, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

42. Secondary Outcome: Subjective Number of Awakenings, Per Post-sleep Questionnaire (Nights 29-30).
Description: as for outcome 40
Time Frame: Nights 29-30
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Number of awakenings per night
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 128 | 130
Number of awakenings per night | 2.8 (0.12) | 2.5 (0.12)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.097, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

43. Secondary Outcome: Subjective Number of Awakenings, Per Post-sleep Questionnaire (Week 2).
Description: The Subjective Number of Awakenings weekly average was the mean of the daily Post-Sleep Questionnaire for the 7 nights prior to the corresponding Visit and predominantly contained data from the natural "home" setting.
Time Frame: Week 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 124 | 127
scores on a scale | 2.2 (0.08) | 2.0 (0.08)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.028, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

44. Secondary Outcome: Subjective Number of Awakenings, Per Post-sleep Questionnaire (Week 4).
Description: as for outcome 43
Time Frame: Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 125 | 127
scores on a scale | 2.2 (0.08) | 1.8 (0.08)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

45. Secondary Outcome: Subjective Number of Awakenings, Per Post-sleep Questionnaire (Week 5).
Description: as for outcome 43
Time Frame: Week 5
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Number analyzed (Participants) | 125 | 127
scores on a scale | 2.3 (0.09) | 2.1 (0.09)
Statistical Analysis 1: Comparison: Placebo QD vs Ramelteon 4 mg QD; Test type: Superiority or Other; p = 0.111, ANCOVA — [p-value comment as in outcome 15, analysis 1]; LS means are from an ANCOVA model with effects for treatment and pooled center, with Baseline as a covariate

ADVERSE EVENTS:
Description: No Serious Adverse Events Reported.
Arm/Group | Placebo QD | Ramelteon 4 mg QD
Serious Adverse Events (participants affected / at risk) | 0/129 | 0/130
Other Adverse Events (participants affected / at risk) | 34/129 | 35/130
OTHER ADVERSE EVENTS (reported when occurring in more than 0.4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD (N=129) | Ramelteon 4 mg QD (N=130)
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Eye Pain (Eye disorders) | 0 | 1
Visual disturbance (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 1 | 2
Pyrexia (Gastrointestinal disorders) | 1 | 1
Inflammation (General disorders) | 0 | 1
Irritability (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 7 | 2
Bronchitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infections (Infections and infestations) | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 3
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Lymphocyte count increased (Investigations) | 1 | 0
Neutrophil count increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Metabolism and nutrition disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 10 | 9
Somnolence (Nervous system disorders) | 1 | 6
Dizziness (Nervous system disorders) | 2 | 2
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Post-traumatic headache (Nervous system disorders) | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 1
Early morning awakenings (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release; such communications can be embargoed for a period up to 150 days to permit actions necessary to preserve sponsor's intellectual property. Sponsor can request changes to the results communication only for the purpose of removing non study related information that is proprietary and confidential to sponsor. Sponsor can require delay of a results communication until the study has been completed at all participating sites.